CLINICAL TRIAL: NCT06227377
Title: A Phase 1 Trial Evaluating the Safety, Tolerability, PK, and Efficacy of QTX3034 in Patients With Solid Tumors With KRASG12D Mutation
Brief Title: QTX3034 in Patients With KRAS G12D Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Quanta Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QTX3034-001
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1a: QTX3034 monotherapy dose-escalation (Experimental): QTX3034 will be administered at protocol defined dose based on cohort assignment
  Interventions: Drug: QTX3034
- Part 1b: QTX3034 combination with cetuximab dose-escalation (Experimental): QTX3034 will be administered at protocol defined dose in combination with cetuximab based on cohort assignment
  Interventions: Drug: QTX3034; Combination Product: Cetuximab
- Part 2: QTX3034 monotherapy dose-expansion (Experimental): QTX3034 will be administered at protocol defined dose in combination with cetuximab based on cohort assignment
  Interventions: Drug: QTX3034
- Part 3: QTX3034 combination with cetuximab dose-expansion (Experimental): QTX3034 will be administered at protocol defined dose in combination with cetuximab based on cohort assignment
  Interventions: Drug: QTX3034; Combination Product: Cetuximab

INTERVENTIONS:
Drug: QTX3034 — QTX3034 will be administered at protocol defined dose
Combination Product: Cetuximab — Cetuximab will be administered at protocol defined dose.
  Arms: Part 1b: QTX3034 combination with cetuximab dose-escalation; Part 3: QTX3034 combination with cetuximab dose-expansion

SUMMARY:
Phase 1 study to determine the safety and tolerability of QTX3034 as a single agent or in combination with cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented, locally advanced or metastatic malignancy with KRAS G12D mutation identified through molecular testing (NGS- or PCR-based) with a Clinical Laboratory Improvement Amendments-certified (or equivalent) diagnostic
* Part 1: - Advanced solid tumors with at least 1 prior systemic therapy
* Evaluable or Measurable disease per RECIST 1.1.
* Parts 2 and 3: Measurable disease per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate organ function

Exclusion Criteria:

* Prior treatment with a KRAS inhibitor
* Active brain metastases or carcinomatous meningitis
* History of other malignancy within 2 years
* Significant cardiovascular disease
* Disease or disorder that may pose a risk to patient's safety

Other protocol-defined Inclusion/Exclusion Criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | up to 21 days
  DLTs will be defined as the occurrence of any of the toxicities as described in the protocol
Number of participants with Treatment-emergent Adverse Events (TEAEs) | up to 2 years
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug monotherapy and in combination with cetuximab

SECONDARY OUTCOMES:
QTX3034 pharmacokinetic parameters in plasma | up to 2 years
  Plasma concentration data for QTX3034 will be used to evaluate PK parameters such as maximum concentration (Cmax), minimum concentration (Cmin), time to attain Cmax (Tmax), area under the concentration-time curve (AUC), elimination half-life (t1⁄2).
Objective response rate (ORR) | up to 2 years
  The ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) based on RECIST 1.1.
Duration of response (DOR) | up to 2 years
  Duration of response (DoR) is defined as the time between first evidence of objective response and disease progression (as measured by RECIST 1.1) or death, whichever occurs earlier, in subjects who achieve CR or PR.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - UCLA Hematology/Oncology, Los Angeles, California
  - Sarah Cannon Research Institute (SCRI), Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - SCRI- Nashville, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - START San Antonio, LLC, San Antonio, Texas
  - University of Utah, Huntsman Cancer Center, Salt Lake City, Utah
  - NEXT Oncology Virginia, Fairfax, Virginia